CLINICAL TRIAL: NCT01983553
Title: Long-Term Follow-Up of Hospitalized Dengue and Safety in Thai Children Who Were Included in an Efficacy Study of a Tetravalent Dengue Vaccine
Brief Title: Long-Term Study of Hospitalized Dengue & Safety in Thai Children Included in a Tetravalent Dengue Vaccine Efficacy Study
Status: Completed | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: CYD57; U1111-1127-7380 (Other: WHO)
Record Dates: First submitted 2013-11-06; First posted 2013-11-14 (Estimated); Results first posted 2019-07-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Dengue; Dengue Fever; Dengue Hemorrhagic Fever
Keywords: Dengue Virus; Dengue Fever; Dengue Hemorrhagic Fever; CYD Dengue Vaccine
MeSH Terms: conditions — Dengue; Severe Dengue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- CYD Dengue Vaccine Group: Participants who received 3 injections of 0.5 milliliter (mL) CYD dengue vaccine, 1 injection each at 0, 6, and 12 months, subcutaneously in study CYD23, were followed up for safety in this study for 4 years after the 3rd vaccination at Month 12 in CYD23.
- Control Group: Participants who received either 0.5 mL Rabies vaccine (Verorab®) or placebo control, subcutaneously as a first injection on Day 0, placebo for second and third injections at 6 and 12 months, respectively in the study CYD23, were followed up for safety in this study for 4 years after the 3rd vaccination at Month 12 in CYD23.

SUMMARY:
The purpose of this study was to conduct a passive surveillance of hospitalized dengue cases in participants who participated in study CYD23 (NCT00842530).

The Objectives:

* To describe the incidence of virologically-confirmed hospitalized dengue cases.
* To characterize hospitalized dengue cases.
* To evaluate the occurrence of related and fatal serious adverse events (SAEs).

DETAILED DESCRIPTION:
This study was a passive surveillance of hospitalized dengue cases in participants who participated in study CYD23 (NCT00842530) where participants were initially randomized to receive 3 injections of either CYD dengue vaccine or control at 6 month intervals. Any SAE related to a study procedure or related to a previous injection from study CYD23, or any fatal SAEs (even if unrelated) were reported to the Sponsor.

An Independent Data Monitoring Committee (IDMC) was also involved in the regular review of virologically-confirmed hospitalized dengue cases. Any fatal outcome or related SAE were be promptly reviewed by the IDMC.

No study vaccinations were administered.

ELIGIBILITY:
Inclusion Criteria:

* Ongoing participation in study CYD23 at the time of enrolment.
* Assent form was signed and dated by the participant (for participants >= 7 years old), and informed consent form was signed and dated by the parent(s) or another legally accepted representative and by 2 independent witnesses.
* Participant and parent/legally accepted representative were able to attend all scheduled visits to comply with all study procedures.

Exclusion Criteria:

* Planned participation in another dengue clinical trial during the present study
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants in study CYD23 (NCT00842530) who were hospitalized with dengue cases.
Sampling Method: Non-Probability Sample
Enrollment: 3203 (Actual)
Dates: Start 2013-09-10 (Actual); Primary Completion 2016-06-15 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (1):
- Ratchaburi, Muang District, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Forrat R, Dayan GH, DiazGranados CA, Bonaparte M, Laot T, Capeding MR, Sanchez L, Coronel DL, Reynales H, Chansinghakul D, Hadinegoro SRS, Perroud AP, Frago C, Zambrano B, Machabert T, Wu Y, Luedtke A, Price B, Vigne C, Haney O, Savarino SJ, Bouckenooghe A, Noriega F. Analysis of Hospitalized and Severe Dengue Cases Over the 6 years of Follow-up of the Tetravalent Dengue Vaccine (CYD-TDV) Efficacy Trials in Asia and Latin America. Clin Infect Dis. 2021 Sep 15;73(6):1003-1012. doi: 10.1093/cid/ciab288. PMID 33822015
- [Derived] Sridhar S, Luedtke A, Langevin E, Zhu M, Bonaparte M, Machabert T, Savarino S, Zambrano B, Moureau A, Khromava A, Moodie Z, Westling T, Mascarenas C, Frago C, Cortes M, Chansinghakul D, Noriega F, Bouckenooghe A, Chen J, Ng SP, Gilbert PB, Gurunathan S, DiazGranados CA. Effect of Dengue Serostatus on Dengue Vaccine Safety and Efficacy. N Engl J Med. 2018 Jul 26;379(4):327-340. doi: 10.1056/NEJMoa1800820. Epub 2018 Jun 13. PMID 29897841
- [Derived] Hadinegoro SR, Arredondo-Garcia JL, Capeding MR, Deseda C, Chotpitayasunondh T, Dietze R, Muhammad Ismail HI, Reynales H, Limkittikul K, Rivera-Medina DM, Tran HN, Bouckenooghe A, Chansinghakul D, Cortes M, Fanouillere K, Forrat R, Frago C, Gailhardou S, Jackson N, Noriega F, Plennevaux E, Wartel TA, Zambrano B, Saville M; CYD-TDV Dengue Vaccine Working Group. Efficacy and Long-Term Safety of a Dengue Vaccine in Regions of Endemic Disease. N Engl J Med. 2015 Sep 24;373(13):1195-206. doi: 10.1056/NEJMoa1506223. Epub 2015 Jul 27. PMID 26214039
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled in the original study CYD23 (NCT00842530) from 10 September 2013 to 29 November 2013 at 1 clinic center in Thailand.
Pre-assignment Details: Of the 3997 participants who were treated in the original study CYD23, a total of 3203 participants were included in this CYD57 study to continue the 4-year safety follow-up.
Groups:
- CYD Dengue Vaccine Group: Participants who received 3 injections of 0.5 mL CYD dengue vaccine, 1 injection each at 0, 6, and 12 months, subcutaneously in study CYD23, were followed up for safety in this study for 4 years after the 3rd vaccination at Month 12 in CYD23.
- Control Group: Participants who received either 0.5 mL Rabies vaccine (Verorab®) or placebo control, subcutaneously as a first injection on Day 0, placebo for second and third injections at 6 and 12 months, respectively, in the study CYD23, were followed up for safety in this study for 4 years after the 3rd vaccination at Month 12 in CYD23.
Period: Overall Study
Arm/Group | CYD Dengue Vaccine Group | Control Group
Started | 2131 | 1072
Completed | 2131 | 1072
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on Follow-up Analysis Set (FupAS) which included all participants who were included in the study CYD57.
Groups:
- Total: Total of all reporting groups
Arm/Group | CYD Dengue Vaccine Group | Control Group | Total
Number analyzed (Participants) | 2131 | 1072 | 3203
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2131 | 1072 | 3203
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.11 (2.02) | 8.15 (2.06) | 8.13 (2.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1118 | 579 | 1697
  Male | 1013 | 493 | 1506

OUTCOME MEASURES:

1. Primary Outcome: Event Rate Per 100 Participant-years for Hospitalized Virologically-Confirmed Dengue (VCD) Cases Due to Any and Each Serotype Following Vaccination With Either CYD Dengue Vaccine or Placebo in the Previous Study (CYD23)
Description: Event rate per 100 participant-years for hospitalized VCD cases, due to any and each serotype (1, 2, 3 and 4) following vaccination with either CYD Dengue vaccine or Placebo in the previous study (CYD23) were reported.
Time Frame: Year 1 to Year 4 post- 3rd vaccination at Month 12 in CYD23
Population: Analysis was performed on FupAS.
Measure: Number (95% Confidence Interval); unit: Events per 100 participant-years
Groups:
- CYD Dengue Vaccine Group: Participants who received 3 injections of 0.5 mL CYD dengue vaccine, 1 injection each at 0, 6, and 12 months, subcutaneously in the previous study CYD23, were followed up for safety in this study for 4 years after the 3rd vaccination at Month 12 in CYD23.
- Control Group: Participants who received either 0.5 mL Rabies vaccine (Verorab®) or placebo control, subcutaneously as a first injection on Day 0, placebo for second and third injections at 6 and 12 months, respectively, in the previous study CYD23, were followed up for safety in this study for 4 years after the 3rd vaccination at Month 12 in CYD23.
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 2131 | 1072
Events per 100 participant-years
  Any of the 4 Serotypes | 1.0 [0.8 to 1.2] | 1.1 [0.8 to 1.4]
  Serotype 1 | 0.2 [0.2 to 0.4] | 0.3 [0.1 to 0.5]
  Serotype 2 | 0.3 [0.2 to 0.5] | 0.3 [0.1 to 0.5]
  Serotype 3 | 0.2 [0.2 to 0.4] | 0.2 [0.1 to 0.4]
  Serotype 4 | 0.2 [0.1 to 0.3] | 0.3 [0.1 to 0.5]
  Unserotyped | 0.0 [0.0 to 0.0] | 0.1 [0.0 to 0.2]
Statistical Analysis 1: Comparison: CYD Dengue Vaccine Group vs Control Group; Relative risk; Any of the 4 Serotypes; Test type: Other — Relative risk analysis of the event rate per 100 participants during Year 1 to Year 4 for Any of the 4 Serotypes between the CYD Dengue vaccine group and the Control group; Relative Risk = 0.930, 95% CI 2-sided [0.64 to 1.36] — The 95% confidence interval of the relative risk was calculated using the Exact method described by Breslow and Day
Statistical Analysis 2: Comparison: CYD Dengue Vaccine Group vs Control Group; Relative risk; Serotype 1; Test type: Other — Relative risk analysis of the event rate per 100 participants during Year 1 to Year 4 for Serotype 1 between the CYD Dengue vaccine group and the Control group; Relative Risk = 0.960, 95% CI 2-sided [0.44 to 2.21] — The 95% confidence interval of the relative risk was calculated using the Exact method described by Breslow and Day
Statistical Analysis 3: Comparison: CYD Dengue Vaccine Group vs Control Group; Relative risk; Serotype 2; Test type: Other — Relative risk analysis of the event rate per 100 participants during Year 1 to Year 4 for Serotype 2 between the CYD Dengue vaccine group and the Control group; Relative Risk = 1.326, 95% CI 2-sided [0.64 to 2.94] — The 95% confidence interval of the relative risk was calculated using the Exact method described by Breslow and Day
Statistical Analysis 4: Comparison: CYD Dengue Vaccine Group vs Control Group; Relative risk; Serotype 3; Test type: Other — Relative risk analysis of the event rate per 100 participants during Year 1 to Year 4 for Serotype 3 between the CYD Dengue vaccine group and the Control group; Relative Risk = 1.056, 95% CI 2-sided [0.48 to 2.51] — The 95% confidence interval of the relative risk was calculated using the Exact method described by Breslow and Day
Statistical Analysis 5: Comparison: CYD Dengue Vaccine Group vs Control Group; Relative risk; Serotype 4; Test type: Other — Relative risk analysis of the event rate per 100 participants during Year 1 to Year 4 for Serotype 4 between the CYD Dengue vaccine group and the Control group; Relative Risk = 0.629, 95% CI 2-sided [0.27 to 1.47] — The 95% confidence interval of the relative risk was calculated using the Exact method described by Breslow and Day
Statistical Analysis 6: Comparison: CYD Dengue Vaccine Group vs Control Group; Relative risk; Unserotyped; Test type: Other — Relative risk analysis of the event rate per 100 participants during Year 1 to Year 4 for Unserotyped between the CYD Dengue vaccine group and the Control group; Relative Risk = 0.000, 95% CI 2-sided [0.00 to 1.22] — The 95% confidence interval of the relative risk was calculated using the Exact method described by Breslow and Day

2. Primary Outcome: Number of Hospitalized VCD Cases Due to Any and Each Serotype (1, 2, 3 and 4) Following Vaccination With Either CYD Dengue Vaccine or a Placebo in a Previous Study (CYD23)
Description: Cases were defined as the number of participants with at least one hospitalized VCD episode.
Time Frame: Year 1 to Year 4 post- 3rd vaccination at Month 12 in CYD23
Population: Analysis was performed on FupAS.
Measure: Number; unit: Cases
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 2131 | 1072
Cases
  Cases: Any of the 4 Serotypes | 85 | 46
  Cases: Serotype 1 | 21 | 11
  Cases: Serotype 2 | 29 | 11
  Cases: Serotype 3 | 21 | 10
  Cases: Serotype 4 | 15 | 12
  Cases: Unserotyped | 0 | 3

3. Primary Outcome: Number of Episodes of Hospitalized VCD Due to Any and Each Serotype (1, 2, 3 and 4) Following Vaccination With Either CYD Dengue Vaccine or a Placebo in a Previous Study (CYD23)
Description: Episodes were defined as the number of hospitalized VCD episodes.
Time Frame: Year 1 to Year 4 post- 3rd vaccination at Month 12 in CYD23
Population: Analysis was performed on FupAS.
Measure: Number; unit: Episodes
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 2131 | 1072
Episodes
  Episodes: Any of the 4 Serotypes | 85 | 46
  Episodes: Serotype 1 | 21 | 11
  Episodes: Serotype 2 | 29 | 11
  Episodes: Serotype 3 | 21 | 10
  Episodes: Serotype 4 | 15 | 12
  Episodes: Unserotyped | 0 | 3

4. Primary Outcome: Event Rate Per 100 Participant-years for Hospitalized VCD Cases Due to Any and Each Serotype Collected By Age Group (Aged: 4-5; 6-11 Years) Following Vaccination With Either CYD Dengue Vaccine or Placebo in a Previous Study (CYD23)
Description: Event rate per 100 participant-years for hospitalized VCD cases, due to any and each serotype (1, 2, 3 and 4) following vaccination with either CYD Dengue vaccine or Placebo in the previous study (CYD23) were reported. Endpoint values <0.1 were rounded to 0.1.
Time Frame: Year 1 to Year 4 post- 3rd vaccination at Month 12 in CYD23
Population: Analysis was performed on FupAS. Here, "number analyzed" signifies participants with available data for each specified category.
Measure: Number (95% Confidence Interval); unit: Events per 100 participant-years
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 2131 | 1072
Events per 100 participant-years
  4 to 5 Years: Any of the 4 Serotypes: number analyzed (Participants) | 393 | 192
  4 to 5 Years: Any of the 4 Serotypes | 1.7 [1.1 to 2.4] | 1.2 [0.5 to 2.2]
  6 to 11 Years: Any of the 4 Serotypes: number analyzed (Participants) | 1738 | 880
  6 to 11 Years: Any of the 4 Serotypes | 0.8 [0.6 to 1.1] | 1.1 [0.7 to 1.4]
  4 to 5 Years: Serotype 1: number analyzed (Participants) | 393 | 192
  4 to 5 Years: Serotype 1 | 0.6 [0.3 to 1.2] | 0.1 [0.0 to 0.7]
  6 to 11 Years: Serotype 1: number analyzed (Participants) | 1738 | 880
  6 to 11 Years: Serotype 1 | 0.2 [0.1 to 0.3] | 0.3 [0.1 to 0.5]
  4 to 5 Years: Serotype 2: number analyzed (Participants) | 393 | 192
  4 to 5 Years: Serotype 2 | 0.4 [0.1 to 0.8] | 0.1 [0.0 to 0.7]
  6 to 11 Years: Serotype 2: number analyzed (Participants) | 1738 | 880
  6 to 11 Years: Serotype 2 | 0.3 [0.2 to 0.5] | 0.3 [0.1 to 0.5]
  4 to 5 Years: Serotype 3: number analyzed (Participants) | 393 | 192
  4 to 5 Years: Serotype 3 | 0.3 [0.1 to 0.7] | 0.3 [0.0 to 0.9]
  6 to 11 Years: Serotype 3: number analyzed (Participants) | 1738 | 880
  6 to 11 Years: Serotype 3 | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.4]
  4 to 5 Years: Serotype 4: number analyzed (Participants) | 393 | 192
  4 to 5 Years: Serotype 4 | 0.4 [0.1 to 0.8] | 0.4 [0.1 to 1.1]
  6 to 11 Years: Serotype 4: number analyzed (Participants) | 1738 | 880
  6 to 11 Years: Serotype 4 | 0.1 [0.1 to 0.2] | 0.3 [0.1 to 0.5]
  4 to 5 Years: Unserotyped: number analyzed (Participants) | 393 | 192
  4 to 5 Years: Unserotyped | 0.0 [0.0 to 0.2] | 0.3 [0.0 to 0.9]
  6 to 11 Years: Unserotyped: number analyzed (Participants) | 1738 | 880
  6 to 11 Years: Unserotyped | 0.0 [0.0 to 0.1] | 0.1 [0.0 to 0.2]
Statistical Analysis 1: Comparison: CYD Dengue Vaccine Group vs Control Group; Relative Risk; 4 to 5 years; Any Serotype; Test type: Other — Relative risk analysis of the event rate per 100 participants during Year 1 to Year 4 for Any of the 4 Serotypes (4 to 5 years) between the CYD Dengue vaccine group and the Control group. Total number of participants analyzed were 585 instead of 3203; Relative Risk = 1.411, 95% CI 2-sided [0.64 to 3.42] — The 95% confidence interval of the relative risk was calculated using the Exact method described by Breslow and Day
Statistical Analysis 2: Comparison: CYD Dengue Vaccine Group vs Control Group; Relative Risk; 6 to 11 years; Any Serotype; Test type: Other — Relative risk analysis of the event rate per 100 participants during Year 1 to Year 4 for Any of the 4 Serotypes (6 to 11 years) between the CYD Dengue vaccine group and the Control group. Total number of participants analyzed were 2618 instead of 3203; Relative Risk = 0.807, 95% CI 2-sided [0.53 to 1.25] — The 95% confidence interval of the relative risk was calculated using the Exact method described by Breslow and Day
Statistical Analysis 3: Comparison: CYD Dengue Vaccine Group vs Control Group; Relative Risk; 4 to 5 years; Serotype 1; Test type: Other — Relative risk analysis of the event rate per 100 participants during Year 1 to Year 4 for Serotype 1 (4 to 5 years) between the CYD Dengue vaccine group and the Control group. Total number of participants analyzed were 585 instead of 3203; Relative Risk = 4.885, 95% CI 2-sided [0.70 to 212.02] — The 95% confidence interval of the relative risk was calculated using the Exact method described by Breslow and Day
Statistical Analysis 4: Comparison: CYD Dengue Vaccine Group vs Control Group; Relative Risk; 6 to 11 years; Serotype 1; Test type: Other — Relative risk analysis of the event rate per 100 participants during Year 1 to Year 4 for Serotype 1 (6 to 11 years) between the CYD Dengue vaccine group and the Control group. Total number of participants analyzed were 2618 instead of 3203; Relative Risk = 0.557, 95% CI 2-sided [0.21 to 1.46] — The 95% confidence interval of the relative risk was calculated using the Exact method described by Breslow and Day
Statistical Analysis 5: Comparison: CYD Dengue Vaccine Group vs Control Group; Relative Risk; 4 to 5 years; Serotype 2; Test type: Other — Relative risk analysis of the event rate per 100 participants during Year 1 to Year 4 for Serotype 2 (4 to 5 years) between the CYD Dengue vaccine group and the Control group. Total number of participants analyzed were 585 instead of 3203; Relative Risk = 2.931, 95% CI 2-sided [0.36 to 134.83] — The 95% confidence interval of the relative risk was calculated using the Exact method described by Breslow and Day
Statistical Analysis 6: Comparison: CYD Dengue Vaccine Group vs Control Group; Relative Risk; 6 to 11 years; Serotype 2; Test type: Other — Relative risk analysis of the event rate per 100 participants during Year 1 to Year 4 for Serotype 2 (6 to 11 years) between the CYD Dengue vaccine group and the Control group. Total number of participants analyzed were 2618 instead of 3203; Relative Risk = 1.165, 95% CI 2-sided [0.53 to 2.74] — The 95% confidence interval of the relative risk was calculated using the Exact method described by Breslow and Day
Statistical Analysis 7: Comparison: CYD Dengue Vaccine Group vs Control Group; Relative Risk; 4 to 5 years; Serotype 3; Test type: Other — Relative risk analysis of the event rate per 100 participants at Year 1 for Serotype 3 (4 to 5 year) between the CYD Dengue vaccine group and the Control group. Total number of participants analyzed were 585 instead of 3203; Relative Risk = 1.221, 95% CI 2-sided [0.20 to 12.83] — The 95% confidence interval of the relative risk was calculated using the Exact method described by Breslow and Day
Statistical Analysis 8: Comparison: CYD Dengue Vaccine Group vs Control Group; Relative Risk; 6 to 11 years; Serotype 3; Test type: Other — Relative risk analysis of the event rate per 100 participants during Year 1 to Year 4 for Serotype 3 (6 to 11 years) between the CYD Dengue vaccine group and the Control group. Total number of participants analyzed were 2618 instead of 3203; Relative Risk = 1.013, 95% CI 2-sided [0.41 to 2.73] — The 95% confidence interval of the relative risk was calculated using the Exact method described by Breslow and Day
Statistical Analysis 9: Comparison: CYD Dengue Vaccine Group vs Control Group; Relative Risk; 4 to 5 years; Serotype 4; Test type: Other — Relative risk analysis of the event rate per 100 participants during Year 1 to Year 4 for Serotype 4 (4 to 5 years) between the CYD Dengue vaccine group and the Control group. Total number of participants analyzed were 585 instead of 3203; Relative Risk = 0.977, 95% CI 2-sided [0.21 to 6.04] — The 95% confidence interval of the relative risk was calculated using the Exact method described by Breslow and Day
Statistical Analysis 10: Comparison: CYD Dengue Vaccine Group vs Control Group; Relative Risk; 6 to 11 years; Serotype 4; Test type: Other — Relative risk analysis of the event rate per 100 participants during Year 1 to Year 4 for Serotype 4 (6 to 11 years) between the CYD Dengue vaccine group and the Control group. Total number of participants analyzed were 2618 instead of 3203; Relative Risk = 0.506, 95% CI 2-sided [0.18 to 1.44] — The 95% confidence interval of the relative risk was calculated using the Exact method described by Breslow and Day
Statistical Analysis 11: Comparison: CYD Dengue Vaccine Group vs Control Group; Relative Risk; 4 to 5 years; Unserotyped; Test type: Other — Relative risk analysis of the event rate per 100 participants during Year 1 to Year 4 for Unserotyped (4 to 5 years) between the CYD Dengue vaccine group and the Control group. Total number of participants analyzed were 585 instead of 3203; Relative Risk = 0.000, 95% CI 2-sided [0.00 to 2.60] — The 95% confidence interval of the relative risk was calculated using the Exact method described by Breslow and Day
Statistical Analysis 12: Comparison: CYD Dengue Vaccine Group vs Control Group; Relative Risk; 6 to 11 years; Unserotyped; Test type: Other — Relative risk analysis of the event rate per 100 participants during Year 1 to Year 4 for Unserotyped (6 to 11 years) between the CYD Dengue vaccine group and the Control group. Total number of participants analyzed were 2618 instead of 3203; Relative Risk = 0.000, 95% CI 2-sided [0.00 to 19.75] — The 95% confidence interval of the relative risk was calculated using the Exact method described by Breslow and Day

5. Primary Outcome: Number of Hospitalized VCD Cases Due to Any and Each Serotype (1, 2, 3 and 4) Collected By Age Group (Aged: 4-5; 6-11 Years) Following Vaccination With Either CYD Dengue Vaccine or Placebo in a Previous Study (CYD23)
Description: Cases were defined as the number of participants with at least one hospitalized VCD episode.
Time Frame: Year 1 to Year 4 post- 3rd vaccination at Month 12 in CYD23
Population: Analysis was performed on FupAS. Here, "number analyzed" signifies participants with evaluable data for each specified category.
Measure: Number; unit: Cases
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 2131 | 1072
Cases
  4 to 5 years cases: Any of the 4 serotype: number analyzed (Participants) | 393 | 192
  4 to 5 years cases: Any of the 4 serotype | 26 | 9
  6 to 11 years cases: Any of the 4 Serotypes: number analyzed (Participants) | 1738 | 880
  6 to 11 years cases: Any of the 4 Serotypes | 59 | 37
  4 to 5 years cases: Serotype 1: number analyzed (Participants) | 393 | 192
  4 to 5 years cases: Serotype 1 | 10 | 1
  6 to 11 years cases: Serotype 1: number analyzed (Participants) | 1738 | 880
  6 to 11 years cases: Serotype 1 | 11 | 10
  4 to 5 years cases: Serotype 2: number analyzed (Participants) | 393 | 192
  4 to 5 years cases: Serotype 2 | 6 | 1
  6 to 11 years cases: Serotype 2: number analyzed (Participants) | 1738 | 880
  6 to 11 years cases: Serotype 2 | 23 | 10
  4 to 5 years cases: Serotype 3: number analyzed (Participants) | 393 | 192
  4 to 5 years cases: Serotype 3 | 5 | 2
  6 to 11 years cases: Serotype 3: number analyzed (Participants) | 1738 | 880
  6 to 11 years cases: Serotype 3 | 16 | 8
  4 to 5 years cases: Serotype 4: number analyzed (Participants) | 393 | 192
  4 to 5 years cases: Serotype 4 | 6 | 3
  6 to 11 years cases: Serotype 4: number analyzed (Participants) | 1738 | 880
  6 to 11 years cases: Serotype 4 | 9 | 9
  4 to 5 years cases: Unserotyped: number analyzed (Participants) | 393 | 192
  4 to 5 years cases: Unserotyped | 0 | 2
  6 to 11 years cases: Unserotyped: number analyzed (Participants) | 1738 | 880
  6 to 11 years cases: Unserotyped | 0 | 1

6. Primary Outcome: Number of Episodes of Hospitalized VCD Due to Any and Each Serotype (1, 2, 3 and 4) Collected By Age Group (Aged: 4-5; 6-11 Years) Following Vaccination With Either CYD Dengue Vaccine or Placebo in a Previous Study (CYD23)
Description: Episodes were defined as the number of hospitalized VCD episodes.
Time Frame: Year 1 to Year 4 post- 3rd vaccination at Month 12 in CYD23
Population: as for outcome 5
Measure: Number; unit: Episodes
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 2131 | 1072
Episodes
  4 to 5 years episodes: Any of 4 serotype: number analyzed (Participants) | 393 | 192
  4 to 5 years episodes: Any of 4 serotype | 26 | 9
  6 to11 years episodes: Any of 4 Serotypes: number analyzed (Participants) | 1738 | 880
  6 to11 years episodes: Any of 4 Serotypes | 59 | 37
  4 to 5 years episodes: Serotype 1: number analyzed (Participants) | 393 | 192
  4 to 5 years episodes: Serotype 1 | 10 | 1
  6 to 11 years episodes: Serotype 1: number analyzed (Participants) | 1738 | 880
  6 to 11 years episodes: Serotype 1 | 11 | 10
  4 to 5 years episodes: Serotype 2: number analyzed (Participants) | 393 | 192
  4 to 5 years episodes: Serotype 2 | 6 | 1
  6 to 11 years episodes: Serotype 2: number analyzed (Participants) | 1738 | 880
  6 to 11 years episodes: Serotype 2 | 23 | 10
  4 to 5 years episodes: Serotype 3: number analyzed (Participants) | 393 | 192
  4 to 5 years episodes: Serotype 3 | 5 | 2
  6 to 11 years episodes: Serotype 3: number analyzed (Participants) | 1738 | 880
  6 to 11 years episodes: Serotype 3 | 16 | 8
  4 to 5 years episodes: Serotype 4: number analyzed (Participants) | 393 | 192
  4 to 5 years episodes: Serotype 4 | 6 | 3
  6 to 11 years episodes: Serotype 4: number analyzed (Participants) | 1738 | 880
  6 to 11 years episodes: Serotype 4 | 9 | 9
  4 to 5 years episodes: Unserotyped: number analyzed (Participants) | 393 | 192
  4 to 5 years episodes: Unserotyped | 0 | 2
  6 to 11 years episodes: Unserotyped: number analyzed (Participants) | 1738 | 880
  6 to 11 years episodes: Unserotyped | 0 | 1

7. Primary Outcome: Event Rate Per 100 Participant-years for Clinically Severe Hospitalized VCD Cases Due to Any and Each Serotype Following Vaccination With Either CYD Dengue Vaccine or Placebo in a Previous Study (CYD23)
Description: Event rate per 100 participant-years for Clinically Severe hospitalized VCD cases, due to any and each serotype (1, 2, 3 and 4) following vaccination with either CYD Dengue vaccine or Placebo in the previous study (CYD23) were reported. Endpoint values <0.1 were rounded to 0.1.
Time Frame: Year 1 to Year 4 post- 3rd vaccination at Month 12 in CYD23
Population: Analysis was performed on FupAS.
Measure: Number (95% Confidence Interval); unit: Events per 100 participant-years
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 2131 | 1072
Events per 100 participant-years
  Any of the 4 Serotypes | 0.1 [0.0 to 0.2] | 0.1 [0.0 to 0.2]
  Serotype 1 | 0.1 [0.0 to 0.2] | 0.0 [0.0 to 0.1]
  Serotype 2 | 0.1 [0.0 to 0.1] | 0.1 [0.0 to 0.1]
  Serotype 3 | 0.1 [0.0 to 0.1] | 0.0 [0.0 to 0.1]
  Serotype 4 | 0.1 [0.0 to 0.1] | 0.1 [0.0 to 0.2]
  Unserotyped | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.1]

8. Primary Outcome: Number of Clinically Severe Hospitalized VCD Cases Due to Any and Each Serotype (1, 2, 3 and 4) Following Vaccination With CYD Dengue Vaccine or Placebo in a Previous Study (CYD23)
Description: Cases were defined as the number of participants with at least one hospitalized VCD episode.
Time Frame: Year 1 to Year 4 post- 3rd vaccination at Month 12 in CYD23
Population: Analysis was performed on FupAS.
Measure: Number; unit: Cases
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 2131 | 1072
Cases
  Cases: Any of the 4 Serotypes | 8 | 3
  Cases: Serotype 1 | 6 | 0
  Cases: Serotype 2 | 1 | 1
  Cases: Serotype 3 | 1 | 0
  Cases: Serotype 4 | 1 | 2
  Cases: Unserotyped | 0 | 0

9. Primary Outcome: Number of Episodes of Clinically Severe Hospitalized VCD Due to Any and Each Serotype (1, 2, 3 and 4) Following Vaccination With CYD Dengue Vaccine or Placebo in a Previous Study (CYD23)
Description: Episodes were defined as the number of hospitalized VCD episodes.
Time Frame: Year 1 to Year 4 post- 3rd vaccination at Month 12 in CYD23
Population: Analysis was performed on FupAS.
Measure: Number; unit: Episodes
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 2131 | 1072
Episodes
  Episodes: Any of the 4 Serotypes | 8 | 3
  Episodes: Serotype 1 | 6 | 0
  Episodes: Serotype 2 | 1 | 1
  Episodes: Serotype 3 | 1 | 0
  Episodes: Serotype 4 | 1 | 2
  Episodes: Unserotyped | 0 | 0

10. Primary Outcome: Number of Cases of Non-Serotype Specific Dengue Viremia Among Hospitalized VCD Cases Following Vaccination With CYD Dengue Vaccine or Placebo in Previous Study (CYD23)
Description: Cases were defined as the number of participants with at least one non-serotype specific dengue viremia among hospitalized VCD cases.
Time Frame: During Year 1 to Year 4 post 3rd vaccination at Month 12 in CYD23 at each of the following time points: Anytime, 0-3 days, 4-7 days, 0-7 days, After 7 days during the sera sample collection time interval of 14 days
Population: Analysis was performed on FupAS. Here, 'number analyzed' = number of hospitalized VCD episodes in the specified time period.
Measure: Number; unit: Participants
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 2131 | 1072
Participants
  Cases - Anytime | 78 | 42
  Cases - 0-3 days | 25 | 12
  Cases - 4-7 days | 53 | 27
  Cases - 0-7 days | 78 | 39
  Cases - After 7 days | NA — No hospitalized VCD case occurred in this specified time period. | 3

11. Primary Outcome: Non-Serotype Specific Dengue Viremia Among Hospitalized VCD Cases Following Vaccination With CYD Dengue Vaccine or Placebo in Previous Study (CYD23)
Description: Quantified viremia was defined as greater than or equal to (>=) lower limit of quantitation (log10 plaque forming unit [pfu]/mL).
Time Frame: Year 1 to Year 4 post-vaccination after 3rd vaccination at Month 12 in CYD23 at each of the following time points: Anytime, 0-3 days, 4-7 days, 0-7 days, After 7 days during the sample collection time interval of 14 days
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: log10 pfu/mL
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 2131 | 1072
log10 pfu/mL
  Mean Viremia - Anytime | 3.64 (1.17) | 3.38 (1.21)
  Mean Viremia - 0-3 days | 4.35 (1.11) | 3.83 (1.53)
  Mean Viremia - 4-7 days | 3.31 (1.06) | 3.12 (0.957)
  Mean Viremia - 0-7 days | 3.64 (1.17) | 3.34 (1.19)
  Mean Viremia - After 7 days | NA (NA) — No hospitalized VCD case occurred in this specified time period. | 3.88 (1.63)

12. Primary Outcome: Event Rate Per 100 Participant-years for Hospitalized VCD Cases Due to Any and Each Serotype and Meeting World Health Organization (WHO) 1997 Criteria Collected Following Either CYD Dengue Vaccine or Placebo in a Previous Study (CYD23)
Description: Event rate per 100 participant-years for hospitalized VCD cases, due to any and each serotype (1, 2, 3 and 4) following vaccination with either CYD Dengue vaccine or Placebo in the previous study (CYD23) were reported. Endpoint values <0.1 were rounded to 0.1. The WHO criteria were fever, any haemorrhagic manifestations, thrombocytopenia, plasma leakage or pleural effusion and/or ascites and/or hypoalbuminemia. Dengue haemorrhagic fever was graded as Grade I: Fever accompanied by non-specific constitutional symptoms; the only hemorrhagic manifestation is a positive tourniquet test. Grade II: Spontaneous bleeding in addition to the manifestations of Grade I participants, usually in the form of skin and/or other hemorrhages. Grade III: Circulatory failure manifested by rapid and weak pulse, narrowing of pulse pressure (20 mmHg or less) or hypotension, with the presence of cold clammy skin and restlessness. Grade IV: Profound shock with undetectable blood pressure and pulse.
Time Frame: Year 1 to Year 4 post- 3rd vaccination at Month 12 in CYD23
Population: Analysis was performed on FupAS.
Measure: Number (95% Confidence Interval); unit: Events per 100 participant-years
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 2131 | 1072
Events per 100 participant-years
  Any of the 4 Serotypes: Any Grade | 0.1 [0.0 to 0.2] | 0.1 [0.0 to 0.2]
  Any of the 4 Serotypes: Grade I | 0.1 [0.0 to 0.1] | 0.1 [0.0 to 0.2]
  Any of the 4 Serotypes: Grade II | 0.1 [0.0 to 0.1] | 0.1 [0.0 to 0.1]
  Any of the 4 Serotypes: Grade III | 0.1 [0.0 to 0.1] | 0.0 [0.0 to 0.1]
  Any of the 4 Serotypes: Grade IV | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.1]
  Serotype 1: Any Grade | 0.1 [0.0 to 0.1] | 0.0 [0.0 to 0.1]
  Serotype 1: Grade I | 0.1 [0.0 to 0.1] | 0.0 [0.0 to 0.1]
  Serotype 1: Grade II | 0.1 [0.0 to 0.1] | 0.0 [0.0 to 0.1]
  Serotype 1: Grade III | 0.1 [0.0 to 0.1] | 0.0 [0.0 to 0.1]
  Serotype 1: Grade IV | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.1]
  Serotype 2: Any Grade | 0.1 [0.0 to 0.1] | 0.1 [0.0 to 0.1]
  Serotype 2: Grade I | 0.1 [0.0 to 0.1] | 0.1 [0.0 to 0.1]
  Serotype 2: Grade II | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.1]
  Serotype 2: Grade III | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.1]
  Serotype 2: Grade IV | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.1]
  Serotype 3: Any Grade | 0.1 [0.0 to 0.1] | 0.0 [0.0 to 0.1]
  Serotype 3: Grade I | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.1]
  Serotype 3: Grade II | 0.1 [0.0 to 0.1] | 0.0 [0.0 to 0.1]
  Serotype 3 Grade III | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.1]
  Serotype 3: Grade IV | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.1]
  Serotype 4: Any Grade | 0.1 [0.0 to 0.1] | 0.1 [0.0 to 0.2]
  Serotype 4: Grade I | 0.0 [0.0 to 0.0] | 0.1 [0.0 to 0.1]
  Serotype 4: Grade II | 0.1 [0.0 to 0.1] | 0.1 [0.0 to 0.1]
  Serotype 4: Grade III | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.1]
  Serotype 4: Grade IV | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.1]
  Unserotyped: Any Grade | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.1]
  Unserotyped: Grade I | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.1]
  Unserotyped: Grade II | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.1]
  Unserotyped: Grade III | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.1]
  Unserotyped: Grade IV | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.1]
Statistical Analysis 1: Comparison: CYD Dengue Vaccine Group vs Control Group; Relative Risk; Any serotype; Any grade; Test type: Other — Relative risk analysis of the event rate per 100 participants during Year 1 to Year 4 for Any of the 4 Serotypes; Any grade between the CYD Dengue vaccine group and the Control group; Relative Risk = 1.174, 95% CI 2-sided [0.27 to 7.03] — The 95% confidence interval of the relative risk was calculated using the Exact method described by Breslow and Day
Statistical Analysis 2: Comparison: CYD Dengue Vaccine Group vs Control Group; Relative Risk; Any serotype; Grade I; Test type: Other — Relative risk analysis of the event rate per 100 participants during Year 1 to Year 4 for Any of the 4 Serotypes; Grade I between the CYD Dengue vaccine group and the Control group; Relative Risk = 0.252, 95% CI 2-sided [0.00 to 4.83] — The 95% confidence interval of the relative risk was calculated using the Exact method described by Breslow and Day
Statistical Analysis 3: Comparison: CYD Dengue Vaccine Group vs Control Group; Relative Risk; Any serotype; Grade II; Test type: Other — Relative risk analysis of the event rate per 100 participants during Year 1 to Year 4 for Any of the 4 Serotypes Grade II between the CYD Dengue vaccine group and the Control group; Relative Risk = 2.012, 95% CI 2-sided [0.20 to 99.10] — The 95% confidence interval of the relative risk was calculated using the Exact method described by Breslow and Day
Statistical Analysis 4: Comparison: CYD Dengue Vaccine Group vs Control Group; Relative Risk; Serotype 2; Any grade; Test type: Other — Relative risk analysis of the event rate per 100 participants during Year 1 to Year 4 for Serotype 2 Any grade between the CYD Dengue vaccine group and the Control group; Relative Risk = 0.503, 95% CI 2-sided [0.01 to 39.49] — The 95% confidence interval of the relative risk was calculated using the Exact method described by Breslow and Day
Statistical Analysis 5: Comparison: CYD Dengue Vaccine Group vs Control Group; Relative Risk; Serotype 2; Grade I; Test type: Other — Relative risk analysis of the event rate per 100 participants during Year 1 to Year 4 for Serotype 2 Grade I between the CYD Dengue vaccine group and the Control group; Relative Risk = 0.503, 95% CI 2-sided [0.01 to 39.49] — The 95% confidence interval of the relative risk was calculated using the Exact method described by Breslow and Day
Statistical Analysis 6: Comparison: CYD Dengue Vaccine Group vs Control Group; Relative Risk; Serotype 4; Any grade; Test type: Other — Relative risk analysis of the event rate per 100 participants during Year 1 to Year 4 for Serotype 4 Any grade between the CYD Dengue vaccine group and the Control group; Relative Risk = 0.252, 95% CI 2-sided [0.00 to 4.83] — The 95% confidence interval of the relative risk was calculated using the Exact method described by Breslow and Day
Statistical Analysis 7: Comparison: CYD Dengue Vaccine Group vs Control Group; Relative Risk; Serotype 4; Grade I; Test type: Other — Relative risk analysis of the event rate per 100 participants during Year 1 to Year 4 for Serotype 4 Grade I between the CYD Dengue vaccine group and the Control group; Relative Risk = 0.000, 95% CI 2-sided [0.00 to 19.62] — The 95% confidence interval of the relative risk was calculated using the Exact method described by Breslow and Day
Statistical Analysis 8: Comparison: CYD Dengue Vaccine Group vs Control Group; Relative Risk; Serotype 4; Grade II; Test type: Other — Relative risk analysis of the event rate per 100 participants during Year 1 to Year 4 for Serotype 4 Grade II between the CYD Dengue vaccine group and the Control group; Relative Risk = 0.503, 95% CI 2-sided [0.01 to 39.49] — The 95% confidence interval of the relative risk was calculated using the Exact method described by Breslow and Day

13. Primary Outcome: Number of Hospitalized VCD Cases Due to Any and Each Serotype (1, 2, 3 and 4) and Meeting WHO 1997 Criteria Following Vaccination With CYD Dengue Vaccine or Placebo in a Previous Study (CYD23)
Description: Cases were defined as the number of participants with at least one hospitalized VCD episode meeting WHO criteria. The WHO criteria was fever, any haemorrhagic manifestations, thrombocytopenia, plasma leakage or pleural effusion and/or ascites and/or hypoalbuminemia. Dengue hemorrhagic fever was graded as - Grade I: Fever accompanied by non-specific constitutional symptoms; the only hemorrhagic manifestation was a positive tourniquet test. Grade II: Spontaneous bleeding in addition to the manifestations of Grade I participants, usually in the form of skin and/or other hemorrhages. Grade III: Circulatory failure manifested by rapid and weak pulse, narrowing of pulse pressure (20 mmHg or less) or hypotension, with the presence of cold clammy skin and restlessness. Grade IV: Profound shock with undetectable blood pressure and pulse.
Time Frame: Year 1 to Year 4 post- 3rd vaccination at Month 12 in CYD23
Population: Analysis was performed on FupAS.
Measure: Number; unit: Cases
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 2131 | 1072
Cases
  Cases: Any of the 4 Serotypes: Any Grade | 7 | 3
  Cases: Any of the 4 Serotypes: Grade I | 1 | 2
  Cases: Any of the 4 Serotypes: Grade II | 4 | 1
  Cases: Any of the 4 Serotypes: Grade III | 2 | 0
  Cases: Any of the 4 Serotypes: Grade IV | 0 | 0
  Cases: Serotype 1: Any Grade | 5 | 0
  Cases: Serotype 1: Grade I | 1 | 0
  Cases: Serotype 1: Grade II | 2 | 0
  Cases: Serotype 1: Grade III | 2 | 0
  Cases: Serotype 1: Grade IV | 0 | 0
  Cases: Serotype 2: Any Grade | 1 | 1
  Cases: Serotype 2: Grade I | 1 | 1
  Cases: Serotype 2: Grade II | 0 | 0
  Cases: Serotype 2: Grade III | 0 | 0
  Cases: Serotype 2: Grade IV | 0 | 0
  Cases: Serotype 3: Any Grade | 1 | 0
  Cases: Serotype 3: Grade I | 0 | 0
  Cases: Serotype 3: Grade II | 1 | 0
  Cases: Serotype 3: Grade III | 0 | 0
  Cases: Serotype 3: Grade IV | 0 | 0
  Cases: Serotype 4: Any Grade | 1 | 2
  Cases: Serotype 4: Grade I | 0 | 1
  Cases: Serotype 4: Grade II | 1 | 1
  Cases: Serotype 4: Grade III | 0 | 0
  Cases: Serotype 4: Grade IV | 0 | 0
  Cases: Unserotyped: Any Grade | 0 | 0
  Cases: Unserotyped: Grade I | 0 | 0
  Cases: Unserotyped: Grade II | 0 | 0
  Cases: Unserotyped: Grade III | 0 | 0
  Cases: Unserotyped: Grade IV | 0 | 0

14. Primary Outcome: Number of Episodes of Hospitalized VCD Cases Due to Any and Each Serotype (1, 2, 3 and 4) and Meeting WHO 1997 Criteria Following Vaccination With CYD Dengue Vaccine or Placebo in a Previous Study (CYD23)
Description: Episodes were defined as the number of hospitalized virologically confirmed dengue episodes meeting WHO criteria. The WHO criteria was fever, any haemorrhagic manifestations, thrombocytopenia, plasma leakage or pleural effusion and/or ascites and/or hypoalbuminemia. Dengue haemorrhagic fever was graded as Grade I: Fever accompanied by non-specific constitutional symptoms; the only hemorrhagic manifestation is a positive tourniquet test. Grade II: Spontaneous bleeding in addition to the manifestations of Grade I participants, usually in the form of skin and/or other hemorrhages. Grade III: Circulatory failure manifested by rapid and weak pulse, narrowing of pulse pressure (20 mmHg or less) or hypotension, with the presence of cold clammy skin and restlessness. Grade IV: Profound shock with undetectable blood pressure and pulse.
Time Frame: Year 1 to Year 4 post- 3rd vaccination at Month 12 in CYD23
Population: Analysis was performed on FupAS.
Measure: Number; unit: Episodes
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 2131 | 1072
Episodes
  Episodes: Any of the 4 Serotypes: Any Grade | 7 | 3
  Episodes: Any of the 4 Serotypes: Grade I | 1 | 2
  Episodes: Any of the 4 Serotypes: Grade II | 4 | 1
  Episodes: Any of the 4 Serotypes: Grade III | 2 | 0
  Episodes: Any of the 4 Serotypes: Grade IV | 0 | 0
  Episodes: Serotype 1: Any Grade | 5 | 0
  Episodes: Serotype 1: Grade I | 1 | 0
  Episodes: Serotype 1: Grade II | 2 | 0
  Episodes: Serotype 1: Grade III | 2 | 0
  Episodes: Serotype 1: Grade IV | 0 | 0
  Episodes: Serotype 2: Any Grade | 1 | 1
  Episodes: Serotype 2: Grade I | 1 | 1
  Episodes: Serotype 2: Grade II | 0 | 0
  Episodes: Serotype 2: Grade III | 0 | 0
  Episodes: Serotype 2 Grade IV | 0 | 0
  Episodes: Serotype 3: Any Grade | 1 | 0
  Episodes: Serotype 3: Grade I | 0 | 0
  Episodes: Serotype 3: Grade II | 1 | 0
  Episodes: Serotype 3: Grade III | 0 | 0
  Episodes: Serotype 3: Grade IV | 0 | 0
  Episodes: Serotype 4: Any Grade | 1 | 2
  Episodes: Serotype 4: Grade I | 0 | 1
  Episodes: Serotype 4: Grade II | 1 | 1
  Episodes: Serotype 4: Grade III | 0 | 0
  Episodes: Serotype: 4 Grade IV | 0 | 0
  Episodes: Unserotyped: Any Grade | 0 | 0
  Episodes: Unserotyped: Grade I | 0 | 0
  Episodes: Unserotyped: Grade II | 0 | 0
  Episodes: Unserotyped: Grade III | 0 | 0
  Episodes: Unserotyped: Grade IV | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected throughout the study period (Year 1 to Year 4 post- 3rd vaccination at Month 12 in CYD23)
Description: This study involved a passive surveillance of hospitalized dengue cases and related and fatal serious adverse events in participants that participated in a previous study (CYD23). Non-serious adverse event data was not collected since no vaccine was administered in the present study. Analysis was performed on FupAS.
Arm/Group | CYD Dengue Vaccine Group | Control Group
All-Cause Mortality (participants affected / at risk) | 3/2131 | 2/1072
Serious Adverse Events (participants affected / at risk) | 3/2131 | 2/1072
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYD Dengue Vaccine Group (N=2131) | Control Group (N=1072)
Gun-shot wound (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Drowning (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.